CLINICAL TRIAL: NCT04159727
Title: Gut Microbiota Dysbiosis and Translocation Within Patients Suffering From Diseases Associated With Increased Intestinal Barrier Permeability : IBD and Parkinson
Brief Title: Gut Microbiota Dysbiosis and Translocation During IBD and Parkinson
Acronym: Medibiote1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 18-22
Record Dates: First submitted 2019-10-16; First posted 2019-11-12 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2019-11

CONDITIONS: Inflammatory Bowel Diseases; Parkinson Disease
Keywords: gut microbiota; Bacterial translocation
MeSH Terms: conditions — Inflammatory Bowel Diseases; Parkinson Disease | interventions — Defecation; Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBD or PD patients (Experimental): 20 patients suffering from IBD 10 patients suffering from PD
  Interventions: Other: stool and blood analysis
- Asymptomatic subjects (Active Comparator): 30 asymptomatic subjects matched to patients on age, sexe and BMI
  Interventions: Other: stool and blood analysis

INTERVENTIONS:
Other: stool and blood analysis — High throughput sequencing and quantitative PCR

SUMMARY:
Inflammatory bowel diseases (IBD) and Parkinson disease (PD) are complex and multifactorial pathologies. Gut microbiota seems to play an active role. Indeed the digestive microbiota of patients with IBD or PD exhibits different compositions compared with asymptomatic subjects.

Bacterial translocation from gut to blood has been reported.

DETAILED DESCRIPTION:
The investigators designed a case-control study to investigate the digestive microbiota and bacterial translocation during IBD and PD. The investigators want to evaluate gut microbiota bacteria involved in dysbiosis and bacterial translocation during IBD and PD. The investigators want to identify bacterial populations that can serve as biomarkers for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* PD patients : age < or = 60 years
* asymptomatic subjects : no chronic disease
* asymptomatic subjects : no treatment

Exclusion Criteria:

* severe anemia (Hb<7g/L)
* people who don't read french
* pregnant women
* people treated by antibiotic, probiotic or prebiotic during the 2 month before inclusion
* people with any diagnosed or treated pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
16S RNA sequencing in stool sample | 2 years
  16S RNA sequencing to identify species constituting the microbiota in the stool
16S RNA sequencing in blood sample | 2 years
  16S RNA sequencing to identify species constituting the microbiota in the blood
Stool quantification of key bacteria associated with intestinal barrier permeability. | 2 years
  To determine stool rates of Faecalibacterium prausnitzii, Akkermansia muciniphila, Bacteroides fragilis, Clostridium difficile, Mycobacterium avium paratuberculosis and Escherischia coli by qPCR
Blood quantification of key bacteria associated with intestinal barrier permeability. | 2 years
  To determine blood rates of Faecalibacterium prausnitzii, Akkermansia muciniphila, Bacteroides fragilis, Clostridium difficile, Mycobacterium avium paratuberculosis and Escherischia coli by qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Philippe HALFON, MD, PhD, Principal Investigator — Hôpital Européen Marseille
Locations (1):
- European Hospital, Marseille, Bouches-du Rhone, France

IPD SHARING:
Plan to Share IPD: No